CLINICAL TRIAL: NCT04235946
Title: Feasibility Study of an Adapted and Supported Water Polo Program to Reduce Fatigue Related to Cancer and Improve Psychological and Social Recovery in Patients With Breast Cancer Remission
Acronym: AQUA-POLO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: Laboratoire Management Sport Cancer EA 4670 (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Aqua POLO-IPC 2019-028; 2019-A03003-54 (Other: ANSM)
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Cancer Related Fatigue; Breast Cancer
Keywords: cancer related fatigue; adapted physical activity
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, monocentric study, which aims to show that physical activity carried out within a high-level structure and coached by elite trainers contributes to psychological and social recovery and to the reduction of fatigue in patients in remission breast cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- accompanied and adapted water polo program (Experimental): 16 and 20 aqua polo sessions (adapted water polo) over a period of 20 weeks, at the rate of one session per week at the Cercle des Nageurs de Marseille (CNM). They will be divided into 3 cycles imitating the preparation of the season of a high-level athlete: a first cycle intended for physical preparation, a second cycle intended for practical learning (technique and tactics) and the third cycle for preparation of a mini tournament.
  Each session will be organized as follows: 1 hour of training in the water followed by 30 min of "debriefing" as a team or individually with the coach. The announced duration of the session will be 2 hours, transport and changing rooms included.
  Interventions: Other: accompanied and adapted water polo program

INTERVENTIONS:
Other: accompanied and adapted water polo program — Validated questionnaires in French will measure fatigue, quality of life, post-traumatic growth and the coach-athlete relationship. All questionnaires will be administered face to face before the sessions by a member of the social psychology research team.
  The collection of qualitative data (semi-structured interviews) will be carried out by one of the members of the research team in social psychology on three occasions (inclusion, Week 10 and Week 20) in order to assess the psychological variables of interest (quality interpersonal relationships, self-esteem, post-traumatic growth) and their dynamics.
  Physiological variables (weight, fat / lean mass, capacity of the operated arm) will be evaluated monthly. The physical measurement data will be recorded in an electronic case report form

SUMMARY:
The main objective of the study is to assess the feasibility of a coached physical activity program in the form of an accompanied and adapted water polo program by evaluating the interest aroused in patients for this proposal. treatments (number of participants and sessions performed).

DETAILED DESCRIPTION:
Prospective, non-randomized, monocentric study, which aims to show that physical activity carried out within a high-level structure and coached by elite trainers contributes to psychological and social recovery and to the reduction of fatigue in patients in remission breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Woman aged 18 to 65, with a good understanding and good practice of the French language.
2. Having been diagnosed with breast cancer: any type of cancer, any type of treatment. Inclusion from 3 weeks to 3 months after the end of treatment (excluding hormone therapy and immunotherapy) Patients who have undergone surgery may be included from 6 weeks post-operative.
3. Signed consent to participate.
4. Affiliation to a social security scheme or beneficiary of such a scheme.
5. Live within a maximum radius of 40 km around Marseille.
6. Swimming skills (basic level).

Exclusion Criteria:

1. Being undergoing chemotherapy treatment
2. Unacquired healing
3. Metastatic cancers
4. Proven psychological pathology proven according to diagnostic criteria (DSM-V)
5. Pregnant or lactating woman

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2021-12-15 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of maintenance of a high level of adherence to the program of physical activities | 20 WEEKS
  the percentage of patients performing 60% of the scheduled sessions. The proposal to participate in this program will be made by the surgeon, oncologist or radiotherapist.

CONTACTS AND LOCATIONS:
Overall Officials: Monique COHEN, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Cercle des nageurs de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cuvelier S, Goetgheluck-Villaron C, Cohen M, Tallet A, Berline M, Boher JM, Jowett S, Justafre S, Dantin P, Viens P, Calvin S. Aqua polo: Preliminary feasibility and efficacy study of a programme of adapted, supervised water polo to reduce fatigue and improve women's psychological and social recovery after breast cancer treatment: A mixed-methods design. Contemp Clin Trials Commun. 2023 Mar 22;33:101120. doi: 10.1016/j.conctc.2023.101120. eCollection 2023 Jun. PMID 37026030